CLINICAL TRIAL: NCT05852275
Title: O-LIVE: Impact of a Portuguese Olive Oil in Health Biomarkers
Acronym: O-LIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Católica Portuguesa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Project nº 171-CES/UCP
Record Dates: First submitted 2023-04-05; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Adult Healthy Volunteers
Keywords: Olive oil; inflammation; gut microbiota; Mediterranean Diet
MeSH Terms: conditions — Inflammation | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: This project consists of a quasi-experimental clinical study whose target population is healthy, voluntary adults. Participants will be recruited among men and women, aged 18 years or over, healthy, who belong to the community of the University (Portuguese Catholic University - Porto campus) and who do not meet any of the exclusion criteria.
  Individuals will be invited to participate voluntarily in this study, receiving detailed information about the investigation, in order to allow an informed, informed and free decision. Individuals who agree to participate sign an informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olive oil arm (Experimental): Participants will include, in their usual diet, the daily intake of 30 mL of an olive oil rich in polyphenols (intervention group) for 100 days. At the beginning (day 1), in the middle (between days 50 and 60) and at the end of the intervention period (day 100), participants will be evaluated.
  Interventions: Other: Olive-oil

INTERVENTIONS:
Other: Olive-oil — Participants will add to their usual diet a daily intake of 30 mL of an olive oil rich in polyphenols for 3-months (100 days)

SUMMARY:
This research project, approved and funded, is part of a larger project, entitled "Healthy Soil for Food", which completes several work packages, one of which is a clinical research submitted to Ethics Committee entitled "O-LIVE: Impact of olive oil Portuguese in biomarkers of healthy volunteers".

The main objective of this work is to evaluate the impact of ingestion of an olive oil rich in polyphenols on clinical biomarkers and parameters, such as anthropometric measurements, on inflammatory gene expression regulation and on the composition of the intestinal microbiota.

DETAILED DESCRIPTION:
Olive oil is an ancient product that is crucial for social cohesion and for local economies in the Mediterranean region, particularly in Portugal. There is ample evidence on the protective effect of olive oil in cardiovascular disease, diabetes, oncological diseases and neurological degeneration. Furthermore, olive oil has been shown to increase the rate of oxidation, inhibiting lipogenesis and stimulating lipolysis, in addition to affecting the expression of receptors involved in weight regulation and fat use.

These health benefits of olive oil derive from its specific nutritional composition, with monounsaturated fatty acids, polyphenols and phenolic compounds, which act on metabolism, modulation of inflammatory responses and gene expression. But the composition of olive oil can vary considerably depending on the type of cultivation of olive trees, soil management practices, as well as the extraction and technological processes involved in olive oil production.

In this work the investigators will use an olive oil rich in polyphenols (produced in a sustainable and local manner) and evaluate its effect on several important clinical parameters involved in chronic diseases. The investigators anticipate that the results of this work will help support the relationship between consuming higher polyphenol olive oil and improved overall health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Current active infections
* Medications (Antidepressant medication, Antibiotics, anti-inflammatory, Angiotensin Converting Enzyme inhibitors, insulin and oral anti-diabetic medication)
* Dietary supplements (minerals and oligoelements, antioxidants, n-3 polyunsaturated fatty acids, n-6 polyunsaturated fatty acids, n-9 fatty acids)
* Presence of ant chronic/metabolic diseases:
* Diabetes
* Cancer
* Inflammatory diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | Day 1
  Body weight will be assessed using a scale
Body weight | Day 50-60
  Body weight will be assessed using a scale
Body weight | Day 100
  Body weight will be assessed using a scale
Bacterial populations in fecal cultures | Day 1
  Bacterial populations in fecal cultures will be analysed by microbial DNA extraction and quantitative real-time polymerase-chain reaction (PCR) using specific primers.
Bacterial populations in fecal cultures | Day 100
  Bacterial populations in fecal cultures will be analyzed by microbial DNA extraction and quantitative real-time polymerase-chain reaction (PCR) using specific primers.
Inflammatory gene expression | Day 1
  Saliva sample will also be collected for subsequent DNA extraction and application of quantitative real-time PCR to determine the expression of inflammatory genes.
Inflammatory gene expression | Day 100
  Saliva sample will also be collected for subsequent DNA extraction and application of quantitative real-time PCR to determine the expression of inflammatory genes.
Body composition (% of fat mass and % of non-fat mass) | Day 1
  Body composition will be assessed using Body Impedance Analysis (body composition analyser)
Body composition (% of fat mass and % of non-fat mass) | Day 100
  Body composition will be assessed using Body Impedance Analysis (body composition analyser)
Adhesion to mediterranean diet | Day 1
  PREDIMED (PREvencion con Diet MEDiterranea) is a brief 14-item tool able to capture a strong monotonic inverse association between adherence to a good quality dietary pattern (Mediterranean diet) and obesity indexes in a population of adults (doi:10.1371/journal.pone.0043134)
Adhesion to mediterranean diet | Day 50-60
  PREDIMED (PREvencion con Diet MEDiterranea) is a brief 14-item tool able to capture a strong monotonic inverse association between adherence to a good quality dietary pattern (Mediterranean diet) and obesity indexes in a population of adults (doi:10.1371/journal.pone.0043134)
Adhesion to mediterranean diet | Day 100
  PREDIMED (PREvencion con DIeta MEDiterranea) is a brief 14-item tool able to capture a strong monotonic inverse association between adherence to a good quality dietary pattern (Mediterranean diet) and obesity indexes in a population of adults (doi:10.1371/journal.pone.0043134)
Lipid profile serum level | Day 1
  A drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for total cholesterol, HDL, LDL and triacylglycerols
Lipid profile serum level | Day 100
  A drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for total cholesterol, HDL, LDL and triacylglycerols
C-reactive Protein serum level | Day 1
  A drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for PCR levels
C-reactive Protein serum level | Day 100
  A drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for PCR levels
glycated hemoglobin A1c serum levels | Day 1
  drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for levels glycated hemoglobin (ha1c)
glycated hemoglobin A1c serum levels | Day 100
  drop of blood will be analysed for biochemical parameters with point of care technology using a finger prick and analysed for levels glycated hemoglobin (ha1c)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gomes, PhD, Study Director — Universidade Católica Portuguesa
Locations (1):
- Escola Superior de Biotecnologia, Universidade Católica Portuguesa, Porto, Portugal

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT05852275/Prot_SAP_ICF_000.pdf